CLINICAL TRIAL: NCT05528432
Title: ANKLE TRAUMA Diagnostic Value of Ultrasound Compared to Standard Radiography in the Detection of Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Other Study IDs: CE-21-02-21
Record Dates: First submitted 2022-08-30; First posted 2022-09-06 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Fractures Bone
Keywords: Fracture ankle; Fracture foot; Frature metatarsus; Ultrasound; X-ray
MeSH Terms: conditions — Fractures, Bone; Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the diagnostic value of ultrasound performed by a lay experimenter compared to standard radiographic imaging (or standard x-ray) in the detection of fractures in patients with closed acute ankle trauma and positive Ottawa ankle rules

DETAILED DESCRIPTION:
Selection of patients is according to the criteria detailed below. If the patient is deemed eligible for the study, he will be asked to read and sign the informed consent. Besides standard history taking, physical examination and radiographic imaging, a standardized ultrasound examination of the ankle joint will be performed by a lay experimenter.

Care will be provided by the attending physician and, according to "standard of care", treatment decisions will be based on history taking, physical examination and conventional ankle x-ray series. Sonographic results will not be used for this purpose. All ankle x-ray series will be reviewed by a senior resident radiologist.

ELIGIBILITY:
Inclusion Criteria:

Any adult patient with acute ankle trauma

+ one or more criteria of the Ottawa ankle rules :

* Inability to walk 4 steps immediately after the trauma or in the emergency room,
* pain at the level of the internal or external malleolus (the distal 6 cm) or the base of the 5th metatarsal bone.

Exclusion Criteria:

* Any patient under the age of 18 years
* Any patient unable to sign the informed consent
* Skin lesions contraindicating sonography (e.g. open fracture wound, … )
* An unstable patient whose inclusion in the study would delay vital treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient presenting to the emergency services of the CHU Saint Pierre
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value | at inclusion
  Negative predictive value of ultrasound compared to standard radiography in the detection of long bone fractures

SECONDARY OUTCOMES:
Sensitivity | at inclusion
  of ultrasound compared to standard radiography in the detection of long bone fractures
Specificity | at inclusion
  of ultrasound compared to standard radiography in the detection of long bone fractures

CONTACTS AND LOCATIONS:
Overall Officials: Laeticia Vaiana FL Frezals, Médecin, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- FREZALS Laeticia Vaiana, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bozkurt O, Ersel M, Karbek Akarca F, Yalcinli S, Midik S, Kucuk L. The diagnostic accuracy of ultrasonography in determining the reduction success of distal radius fractures. Turk J Emerg Med. 2018 Aug 10;18(3):111-118. doi: 10.1016/j.tjem.2018.04.001. eCollection 2018 Sep. PMID 30191190
- [Derived] Frezals LV, Delafontaine A, Scoubeau H, Sontou R, Moorthamers S, Plumacker A, Plumacker A. Diagnostic value of FAST ankle ultrasound compared to standard radiography for fracture detection in the emergency department by non-radiologist physicians: a monocentric prospective diagnostic cohort study. Eur J Trauma Emerg Surg. 2025 Feb 14;51(1):107. doi: 10.1007/s00068-025-02772-3. PMID 39953135
- See also: Ferràs-Tarragó, J., Antequera-Cano, J.M., Català-de-las-Marinas, J. et al. Ankle torque-related fractures and its echo-fast diagnosis protocol. Eur J Trauma Emerg Surg 46, 801-805 (2020) — https://doi.org/10.1007/s00068-018-01069-y
- See also: Doherty, C., Delahunt, E., Caulfield, B. et al. The Incidence and Prevalence of Ankle Sprain Injury: A Systematic Review and Meta-Analysis of Prospective Epidemiological Studies. Sports Med 44, 123-140 (2014) — https://doi.org/10.1007/s40279-013-0102-5
- See also: Champagne N, Eadie L, Regan L, Wilson P. The effectiveness of ultrasound in the detection of fractures in adults with suspected upper or lower limb injury: a systematic review and subgroup meta-analysis. BMC Emergency Medicine 2019;19 — https://doi.org/10.1186/s12873-019-0226-5
- See also: Nelson BP, Chason K. Use of ultrasound by emergency medical services: a review. International Journal of Emergency Medicine 2008 12;1(4):253-259 — https://doi.org/10.1186/s12873-019-0226-5